CLINICAL TRIAL: NCT04174430
Title: Clinical and Paraclinical Characteristics of Severe Bronchiolitis in Children From 2 Months to 12 Months at the Children's Hospital 1 in Ho Chi Minh City - Vietnam
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, LAN HUYNH CHI, Pediatric Resident, Clinical Physician, Respiratory Department, Children Hospital N01, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: IRB00010193
Record Dates: First submitted 2019-11-16; First posted 2019-11-22 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Epidemiological, Clinical, Paraclinical Characterictics of Severe Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mild to moderate bronchiolitis: Bronchiolistis patients without Prematurity (gestational age ≤36 weeks), Low birth weight, Age less than 12 weeks, Chronic pulmonary disease, particularly bronchopulmonary dysplasia (also known as chronic lung disease), Anatomic defects of the airways, Hemodynamically significant congenital heart disease, Immunodeficiency and Neurologic disease
  Interventions: Biological: severe bronchiolitis

INTERVENTIONS:
Biological: severe bronchiolitis — Prematurity (gestational age ≤36 weeks), Low birth weight, Age less than 12 weeks,Chronic pulmonary disease, particularly bronchopulmonary dysplasia (also known as chronic lung disease), Anatomic defects of the airways, Hemodynamically significant congenital heart disease, Immunodeficiency, Neurologic disease

SUMMARY:
Goal: The aim of this study is to determine the epidemiological, clinical, paraclinical characteristics and treatment of severe bronchiolitis at the Children Hospital N01 in 2001-2002.

Materials and method: in this cross-sectional study, specimens of 51 patients with severe bronchiolitis at the Children Hospital N01 from March, 1 st 2001 to February, 28th 2002 are described and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* children younger from 2-12 months present fever (usually ≤38.3ºC [101ºF]) ,cough, and respiratory distress (eg, increased respiratory rate, retractions, wheezing, crackles)
* preceded by a one- to three-day history of upper respiratory tract symptoms (eg, nasal congestion and/or discharge) ]
* Respiratory distress.

Exclusion Criteria:

* refusal to give informed consent
* mucus sample Barlett <=0

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children younger from 2-12 months are diagnosed broncholitis in children hospital 1
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Severe bronchiolitis at the Children Hospital N01 | 2 years
  Bronchiolitis in infants with:
  * Preterm birth : gestational age < 37 weeks
  * Respiratory failure:
    * Irritable condition
    * Breath rate > 50 per minute
    * Hypoxiemia: SpO2 < 94%
  * Poor feeding
  * Hemodynamically significant congenital heart disease (congennital heart failure, moderate to severe pulmonary hypertension or cyanotic heart disease)

CONTACTS AND LOCATIONS:
Overall Officials: Thinh Tan Nguyen, professor, Study Director — HoChiMinh Medical University
Locations (1):
- Respiratory, Ho Chi Minh City, District 10, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
not yet

REFERENCES:
- [Result] Saez-Lopez E, Cristovao P, Costa I, Pechirra P, Conde P, Guiomar R; Portuguese Laboratory Network for the Diagnosis of Influenza Infection; Peres MJ, Viseu R, Lopes P, Soares V, Vale F, Fonseca P, Freitas L, Alves J, Pessanha MA, Toscano C, Mota-Vieira L, Veloso RC, Corte-Real R, Branquinho P, Pereira-Vaz J, Rodrigues F, Cunha M, Martins L, Mota P, Couto AR, Bruges-Armas J, Almeida S, Rodrigues D. Epidemiology and genetic variability of respiratory syncytial virus in Portugal, 2014-2018. J Clin Virol. 2019 Dec;121:104200. doi: 10.1016/j.jcv.2019.104200. Epub 2019 Oct 10. PMID 31707201
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/31707201